CLINICAL TRIAL: NCT04480281
Title: Intravenous Lidocaine Reduces Pain Scores and Opioid Consumption in Open Lung Resection Surgery: A Prospective Randomized Double-Blind Controlled Trial
Brief Title: Intravenous Lidocaine in Open Lung Resection Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Afrida Gergess, Anesthesiologist specialized in cardiovascular and thoracic surgery, Saint-Joseph University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEHDF 972
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Lidocaine; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine Group (Active Comparator): Bolus of lidocaine 1% 1.5mg/kg at the induction of general anesthesia followed by a continuous infusion of lidocaine 1% 2mg/kg/h just before surgical incision and continued until 24h after the surgery
  Interventions: Drug: Lidocaine Iv
- Placebo Group (Placebo Comparator): Equal bolus volume of normal saline solution at induction, and then a continuous infusion started before surgical incision and maintained up until 24h postoperatively
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Lidocaine Iv — Patients in the Lidocaine group received a bolus of lidocaine 1% 1.5mg/kg at the induction of general anesthesia followed by a continuous infusion of lidocaine 1% 2mg/kg/h just before surgical incision and continued until 24h after the surgery
  Arms: Lidocaine Group
Drug: Normal Saline — Patients in Group Placebo received an equal bolus volume of normal saline solution at induction, and then a continuous infusion started before surgical incision and maintained up until 24h postoperatively
  Arms: Placebo Group

SUMMARY:
Management of postoperative pain in 2020 remains a challenge for anesthesiologists in the perioperative period. Lidocaine is an amide local anesthetic, it is one of the oldest adjuvant analgesics and is known to possess analgesic, anti-hyperalgesic and anti-inflammatory properties. Lidocaine is proven to be as effective as epidural analgesia in colorectal surgery.

However, no study has evaluated the effect of a continuous lidocaine infusion for open lung resection in the post-operative period. The present study aims to evaluate the influence of IV lidocaine given during and 24 hours after surgery, on pain scores, opioid consumption, and possible benefits on patient outcome via the opioid-sparing effect in open thoracic surgery

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists (ASA) scores of I, II or III.
* Left or right posterolateral thoracotomy with postoperative monitoring in the intensive care unit (ICU) for at least 24 hours (h).

Exclusion Criteria:

* patient's refusal to participate
* ASA score of IV or higher
* severe hepatic or renal insufficiency
* allergy to lidocaine, morphine or NSAIDs
* cardiac arrhythmias or
* epilepsy,
* delayed extubation for more than 2 h postoperatively
* urgent surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Opioid consumption in the post operative period | Doses were measured for twenty four hours in the post operative period
  Total dose of morphine in the post operative period is measured for patients in both arms
Pain scores at rest and at cough | Measurements were made for 24 hours in the post operative period
  Analogue visual scale ( a 10cm scale , zero representing no pain and 10 representing the worst imaginable pain)) was used to measure pain scores for each patient at rest and at cough

SECONDARY OUTCOMES:
Pulmonary complications | Measurements were recorded for 24 hours in the post operative period
  Arterial partial carbon dioxide pressure (PCO2) measurements were recorded for patients in both arms

CONTACTS AND LOCATIONS:
Locations (1):
- Hotel Dieu de France, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swenson BR, Gottschalk A, Wells LT, Rowlingson JC, Thompson PW, Barclay M, Sawyer RG, Friel CM, Foley E, Durieux ME. Intravenous lidocaine is as effective as epidural bupivacaine in reducing ileus duration, hospital stay, and pain after open colon resection: a randomized clinical trial. Reg Anesth Pain Med. 2010 Jul-Aug;35(4):370-6. doi: 10.1097/AAP.0b013e3181e8d5da. PMID 20588151
- [Result] Cui W, Li Y, Li S, Wang R, Li J. Systemic administration of lidocaine reduces morphine requirements and postoperative pain of patients undergoing thoracic surgery after propofol-remifentanil-based anaesthesia. Eur J Anaesthesiol. 2010 Jan;27(1):41-6. doi: 10.1097/EJA.0b013e32832d5426. PMID 19478674